CLINICAL TRIAL: NCT01075412
Title: 'F-18 Fluorothymidine ([18F]FLT) PET Imaging for Early Evaluation of Response to Chemoradiation Therapy in Patients With Cervical Cancer
Brief Title: FLT PET Imaging for Cervical Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was closed and reopened as NCT01717391
Sponsor: University of Iowa (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sarah McGuire, Assistant Professor of Radiation Oncology, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200906786
Record Dates: First submitted 2010-02-23; First posted 2010-02-25 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Positron-Emission Tomography; Radiotherapy, Intensity-Modulated
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 2 (Experimental): Receives fourth [F18]Fluorothymidine (FLT) PET scan after 20 fractions of radiation therapy.
  Interventions: Drug: [F18]Fluorothymidine
- Group 1 (Experimental): Receives fourth [F18]Fluorothymidine (FLT) PET scan after 15 fractions of radiation therapy.
  Interventions: Drug: [F18]Fluorothymidine

INTERVENTIONS:
Drug: [F18]Fluorothymidine — FLT PET scan 5 mCi (+/- 10%)
  Other Names: FLT

SUMMARY:
Our primary hypothesis is that [18F]FLT PET can identify active bone marrow in addition to metabolically active tumor.

This trial will use FLT-PET imaging to define areas of active bone marrow in the pelvis. The radiation plan is then designed to spare that area, in hopes of keeping the bone marrow active during therapy. Bone marrow and tumor activity will be monitored using a sequence of FLT PET scans during the course of chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
Subjects will undergo a total of up to 5 FLT PET scans.

Subjects are randomized between two groups to reduce radiation exposure from the FLT PET scans. If bone marrow activity is not identified in one scan, further scans are cancelled until the 1-month follow up scan. This is not a randomization to compare therapeutic efficacy between two study arms. Data will be pooled for analysis as pre-specified in the study's statistical plan.

Group 1 has FLT PET scans pretreatment, after 5 radiation treatments, after 10 radiation treatments, after 15 radiation treatments, and then 1 month after completing radiation therapy.

Group 2 has FLT PET scans pretreatment, after 5 radiation treatments, after 10 radiation treatments, after 20 radiation treatments, and then 1 month after completing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Histologically confirmed stage IB2, IIA, IIB, IIIB, and IVA squamous cell carcinoma of the cervix.
* Scheduled to receive chemo-radiation for oncologic treatment.
* Karnofsky of at least 60 at time of screening
* Life expectancy of at least 6 months.
* Leukocytes at least 3,000/microL
* absolute neutrophil count at least 1,500/microL
* platelets at least 100,000/microL
* total bilirubin at maximum 1.0 mg/dL (UIHC limit of normal)
* either ALT or AST less than 2.5 times the upper limit of normal
* creatinine less than 1.5 times the upper limit of normal
* non-pregnant, non-nursing, willing to use contraception

Exclusion Criteria:

* oncology research protocol requiring full pelvic radiation (i.e., 4-field box technique) or experimental chemotherapy
* uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
* subjects taking nucleoside analog medications such as those used as antiretroviral agents.
* patients who have undergone hysterectomy or will have a hysterectomy as part of their cancer therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Graham, Ph.D., M.D., Study Director — University of Iowa; Sarah McGuire, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Yes, data will be shared utilizing clinicaltrials.gov results

REFERENCES:
- [Background] McGuire SM, Menda Y, Ponto LL, Gross B, Juweid M, Bayouth JE. A methodology for incorporating functional bone marrow sparing in IMRT planning for pelvic radiation therapy. Radiother Oncol. 2011 Apr;99(1):49-54. doi: 10.1016/j.radonc.2011.01.025. Epub 2011 Mar 22. PMID 21397965
- [Background] McGuire SM, Menda Y, Boles Ponto LL, Gross B, Buatti J, Bayouth JE. 3'-deoxy-3'-[(1)(8)F]fluorothymidine PET quantification of bone marrow response to radiation dose. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):888-93. doi: 10.1016/j.ijrobp.2010.12.009. Epub 2011 Feb 6. PMID 21300484
- [Background] Menda Y, Ponto LL, Dornfeld KJ, Tewson TJ, Watkins GL, Gupta AK, Anderson C, McGuire S, Schultz MK, Sunderland JJ, Graham MM, Buatti JM. Investigation of the pharmacokinetics of 3'-deoxy-3'-[18F]fluorothymidine uptake in the bone marrow before and early after initiation of chemoradiation therapy in head and neck cancer. Nucl Med Biol. 2010 May;37(4):433-8. doi: 10.1016/j.nucmedbio.2010.02.005. PMID 20447554
- [Result] McGuire SM, Bhatia SK, Sun W, Jacobson GM, Menda Y, Ponto LL, Smith BJ, Gross BA, Bayouth JE, Sunderland JJ, Graham MM, Buatti JM. Using [(18)F]Fluorothymidine Imaged With Positron Emission Tomography to Quantify and Reduce Hematologic Toxicity Due to Chemoradiation Therapy for Pelvic Cancer Patients. Int J Radiat Oncol Biol Phys. 2016 Sep 1;96(1):228-39. doi: 10.1016/j.ijrobp.2016.04.009. Epub 2016 Apr 19. PMID 27319286
- [Result] McGuire SM, Menda Y, Ponto LLB, Gross B, TenNapel M, Smith BJ, Bayouth JE. Spatial mapping of functional pelvic bone marrow using FLT PET. J Appl Clin Med Phys. 2014 Jul 8;15(4):129-136. doi: 10.1120/jacmp.v15i4.4780. PMID 25207403

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Scheduled to receive the fourth [F18]Fluorothymidine (FLT) PET scan after 15 fractions of radiation therapy. If no bone marrow uptake is seen at the second or third FLT PET scan, this scan is omitted to reduce radiation risk.
  [F18]Fluorothymidine: FLT PET scan 5 mCi (+/- 10%)
- Group 2: Receives fourth [F18]Fluorothymidine (FLT) PET scan after 20 fractions of radiation therapy. If no bone marrow uptake is seen at the second or third FLT PET scan, this scan is omitted to reduce radiation risk.
  [F18]Fluorothymidine: FLT PET scan 5 mCi (+/- 10%)
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 4 | 2
Completed | 4 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Difference From Baseline IMRT Plan (%)
Description: The difference in volume of bone marrow receiving radiation using a bone-marrow-sparing radiation plan compared to a standard radiation plan (IMRT), expressed as a percentage. Both plans are patient-specific. Bone-marrow is identified using the baseline FLT PET/CT obtained pre-imaging. Active bone marrow is considered to have an uptake value (SUV) of 2, 3, or 4. The standard IMRT plan was created using the criteria of the National Cancer Institute's Radiation Therapy Oncology Group study RTOG-0418. Radiation dose bins evaluated are 5 Gray, 10 Gray, 20 Gray, and 30 Gray. The change in dose to tumor is also provided. A negative value indicates that more bone marrow or tissue was spared using the bone-marrow sparing plan.
Time Frame: Baseline (pre-treatment)
Population: Participants who received an FLT PET/CT during radiation simulation and did not withdraw from study participation. Groups 1 and 2 were combined as pre-specified in the study protocol, as the groups were separated only to reduce radiation risk from FLT PET imaging (and not for therapeutic comparison).
Measure: Mean (Standard Deviation); unit: Percent difference (%)
Groups:
- All Participants: The outcome measure is evaluated by including study participants from both groups.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Percent difference (%)
  % difference, volume receiving 5 Gray | -8.5 (6.0)
  % difference, volume receiving 10 Gray | -11.7 (7.3)
  % difference, volume receiving 20 Gray | -15.8 (3.8)
  % difference, volume receiving 30 Gray | -16.5 (12.6)
  % difference, dose to target (tumor) volume | -0.2 (0.1)

2. Secondary Outcome: Chemotherapy Compliance
Description: The number of participants who missed at least one prescribed chemotherapy administration due to low blood counts.
Time Frame: post-treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 5
Participants
  Received all chemotherapy as precscribed | 4
  Missed 1 cycle of chemotherapy | 1

3. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for White Blood Cell Counts
Description: White blood cell counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured weekly during combined chemotherapy and radiation therapy treatment and then once at 30 day follow-up and at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, and 30 days post treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 5
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 5
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 5
  Therapy, week 1: CTCAE grade 1 | 0
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 4
  Therapy, week 2: CTCAE grade 1 | 1
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 0
  Therapy, week 2: CTCAE grade 4 (most severe) | 0
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 3
  Therapy, week 3: CTCAE grade 1 | 0
  Therapy, week 3: CTCAE grade 2 | 2
  Therapy, week 3: CTCAE grade 3 | 0
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 0
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 3
  Therapy, week 4: CTCAE grade 1 | 0
  Therapy, week 4: CTCAE grade 2 | 2
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 0
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 2
  Therapy, week 5: CTCAE grade 1 | 0
  Therapy, week 5: CTCAE grade 2 | 1
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 2
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 1
  30 days post-therapy: CTCAE grade 1 | 0
  30 days post-therapy: CTCAE grade 2 | 1
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 3

4. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Platelet Counts.
Description: Platelet cell counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, and 30 days post treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 5
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 5
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 5
  Therapy, week 1: CTCAE grade 1 | 0
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 4
  Therapy, week 2: CTCAE grade 1 | 1
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 0
  Therapy, week 2: CTCAE grade 4 (most severe) | 0
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 3
  Therapy, week 3: CTCAE grade 1 | 2
  Therapy, week 3: CTCAE grade 2 | 0
  Therapy, week 3: CTCAE grade 3 | 0
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 0
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 2
  Therapy, week 4: CTCAE grade 1 | 3
  Therapy, week 4: CTCAE grade 2 | 0
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 0
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 1
  Therapy, week 5: CTCAE grade 1 | 2
  Therapy, week 5: CTCAE grade 2 | 0
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 2
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 2
  30 days post-therapy: CTCAE grade 1 | 0
  30 days post-therapy: CTCAE grade 2 | 0
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 3

5. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Absolute Neutrophil Counts (ANCs)
Description: Absolute neutrophil counts (ANCs) measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up.
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, and 30 days post treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 5
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 5
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 5
  Therapy, week 1: CTCAE grade 1 | 0
  Therapy, week 1: CTCAE grade 2 | 0
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 5
  Therapy, week 2: CTCAE grade 1 | 0
  Therapy, week 2: CTCAE grade 2 | 0
  Therapy, week 2: CTCAE grade 3 | 0
  Therapy, week 2: CTCAE grade 4 (most severe) | 0
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 3
  Therapy, week 3: CTCAE grade 1 | 1
  Therapy, week 3: CTCAE grade 2 | 1
  Therapy, week 3: CTCAE grade 3 | 0
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 0
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 3
  Therapy, week 4: CTCAE grade 1 | 1
  Therapy, week 4: CTCAE grade 2 | 1
  Therapy, week 4: CTCAE grade 3 | 0
  Therapy, week 4: CTCAE grade 4 (most severe) | 0
  Therapy, week 4: Not assessed (test omitted) | 0
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 2
  Therapy, week 5: CTCAE grade 1 | 0
  Therapy, week 5: CTCAE grade 2 | 1
  Therapy, week 5: CTCAE grade 3 | 0
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 2
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 1
  30 days post-therapy: CTCAE grade 1 | 1
  30 days post-therapy: CTCAE grade 2 | 0
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 3

6. Secondary Outcome: Number of Participants With Standardized Toxicity Severity Grades for Decreased Lymphocyte Counts.
Description: Lymphocyte counts measurements expressed in standardized toxicity severity grades (Common Terminology Criteria for Adverse Events, v4.03) measured once weekly during combined chemotherapy and radiation therapy, then once at 30 day follow-up, and once at 1 year follow-up
Time Frame: baseline, weekly during radiation treatment for up to 5 weeks, and 30 days post treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 5
Participants
  Baseline (pre-treatment): CTCAE grade 0 (no toxicity) | 5
  Baseline (pre-treatment): CTCAE grade 1 | 0
  Baseline (pre-treatment): CTCAE grade 2 | 0
  Baseline (pre-treatment): CTCAE grade 3 | 0
  Baseline (pre-treatment): CTCAE grade 4 (most severe) | 0
  Baseline (pre-treatment): Not assessed (test omitted) | 0
  Therapy, week 1: CTCAE grade 0 (no toxicity) | 2
  Therapy, week 1: CTCAE grade 1 | 1
  Therapy, week 1: CTCAE grade 2 | 2
  Therapy, week 1: CTCAE grade 3 | 0
  Therapy, week 1: CTCAE grade 4 (most severe) | 0
  Therapy, week 1: Not assessed (test omitted) | 0
  Therapy, week 2: CTCAE grade 0 (no toxicity) | 1
  Therapy, week 2: CTCAE grade 1 | 1
  Therapy, week 2: CTCAE grade 2 | 1
  Therapy, week 2: CTCAE grade 3 | 1
  Therapy, week 2: CTCAE grade 4 (most severe) | 1
  Therapy, week 2: Not assessed (test omitted) | 0
  Therapy, week 3: CTCAE grade 0 (no toxicity) | 0
  Therapy, week 3: CTCAE grade 1 | 0
  Therapy, week 3: CTCAE grade 2 | 1
  Therapy, week 3: CTCAE grade 3 | 4
  Therapy, week 3: CTCAE grade 4 (most severe) | 0
  Therapy, week 3: Not assessed (test omitted) | 0
  Therapy, week 4: CTCAE grade 0 (no toxicity) | 0
  Therapy, week 4: CTCAE grade 1 | 0
  Therapy, week 4: CTCAE grade 2 | 1
  Therapy, week 4: CTCAE grade 3 | 3
  Therapy, week 4: CTCAE grade 4 (most severe) | 1
  Therapy, week 4: Not assessed (test omitted) | 0
  Therapy, week 5: CTCAE grade 0 (no toxicity) | 0
  Therapy, week 5: CTCAE grade 1 | 0
  Therapy, week 5: CTCAE grade 2 | 2
  Therapy, week 5: CTCAE grade 3 | 1
  Therapy, week 5: CTCAE grade 4 (most severe) | 0
  Therapy, week 5: Not assessed (test omitted) | 2
  30 days post-therapy: CTCAE grade 0 (no toxicity) | 1
  30 days post-therapy: CTCAE grade 1 | 0
  30 days post-therapy: CTCAE grade 2 | 1
  30 days post-therapy: CTCAE grade 3 | 0
  30 days post-therapy: CTCAE grade 4 (most severe) | 0
  30 days post-therapy: Not assessed (test omitted) | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of FLT injection through 24 hours post-injection.
Description: The medical chart was reviewed for possible adverse events post-FLT administration; this is considered non-systematic. The participant was contacted by a licensed healthcare provider to assess for adverse events - this was a systematic approach.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

LIMITATIONS AND CAVEATS:
The results of this pilot study were merged with NCT01717391 for analysis and resultant publication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes